CLINICAL TRIAL: NCT00007670
Title: CSP #428 - Treatment of Seizures in the Elderly Population
Brief Title: Does Gabapentin and Lamotriginel Have Significantly Fewer Side-effects While Providing Equal or Better Seizure Control Than the Current Drug Choice, Carbamazepine, for the Treatment of Seizures in the Elderly.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Parke-Davis (Industry); Glaxo Wellcome (Industry)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 428
Record Dates: First submitted 2000-12-29; First posted 2001-01-04 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Seizures
Keywords: gabapentin; lamotrigine; seizures in the elderly; Carbamazepine
MeSH Terms: conditions — Seizures | interventions — Carbamazepine; Gabapentin; Lamotrigine

INTERVENTIONS:
Drug: Carbamazepine
Drug: Gabapentin
Drug: Lamotrigine

SUMMARY:
New onset epilepsy in the elderly occurs in 45,000-50,000 elderly patients each year. These patients are especially vulnerable to side effects from medications because of changes caused by the aging process and the fact that these patients often have many common diseases for which they are already receiving medications for so that the likelihood of drug interactions is increased. Two new drugs, gabapentin and lamotrigine, have recently been approved by the FDA as antiepileptic drugs. These drugs have demonstrated efficacy in the treatment of partial onset seizures, the most common seizures in the elderly. These new compounds also have favorable side effect profiles and infrequent drug-drug interactions and, therefore, would be expected to be well-tolerated in the elderly.

DETAILED DESCRIPTION:
Primary Hypothesis: The primary hypothesis for this study is that one or both of two newly FDA approved antiepileptic drugs, gabapentin and lamotrigine, will have significantly fewer side-effects while providing equal or possibly better seizure control than the current world-wide drug of choice, carbamazepine, for the treatment of seizures in the elderly.

Secondary Hypotheses: Secondary aims of the study are to determine which of the three drugs being studied (1) has the fewest side-effects, (2) produces the best seizure control, (3) has the least impairment of cognitive function, (4) has the best effect on mood and (5) has the best effect on quality of life.

Intervention: Patients are randomized to carbamazepine, gabapentin or lamotrigine. Target doses are 600mg for carbamazepine (200mg tablets overencapsulated), 1500mg for gabapentin (300mg capsules), and 150mg for lamotrigine (25mg tablets). Carbamazepine and gabapentin patients also receive a placebo tablet while lamotrigine patients also receive a placebo capsule.

Primary Outcomes: The primary outcome measure is retention in the study at 12 months. Major secondary outcomes are seizure frequency during first 12 months, time to first seizure, total scores from Systemic Toxicity and Neurotoxicity Rating Scales, the Mattis Dementia Rating Scale (cognitive function), Hamilton Depression Scale (mood) and SF-36 Health Survey (quality of life).

Study Abstract: New onset epilepsy in the elderly occurs in 45,000-50,000 elderly patients each year. These patients are especially vulnerable to side effects from medications because of changes caused by the aging process and the fact that these patients often have many common diseases for which they are already receiving medications for so that the likelihood of drug interactions is increased. Two new drugs, gabapentin and lamotrigine, have recently been approved by the FDA as antiepileptic drugs. These drugs have demonstrated efficacy in the treatment of partial onset seizures, the most common seizures in the elderly. These new compounds also have favorable side effect profiles and infrequent drug-drug interactions and, therefore, would be expected to be well-tolerated in the elderly. Thus, the primary objective of this study is to evaluate the tolerability and efficacy of these two new antiepileptic drugs individually compared to a standard antiepileptic drug, carbamazepine, in an elderly population (>60 years of age) with new onset, unprovoked epileptic seizures.

The study is a 63-month, randomized, double-blind trial of three antiepileptic drugs: carbamazepine, gabapentin, and lamotrigine. Patient recruitment occured during the first 51 months with each patient being followed for at least one year. There were 593 patients enrolled from 18 VA medical centers. Patients are veterans 60 years of age or older who have new onset, unprovoked seizures of focal onset, with or without secondary generalization. Patients with seizures secondary to toxic-metabolic causes, acute medical or neurological conditions or progressive diseases of the brain such as brain tumors are excluded. A double-dummy design is being employed to preserve the blind. Target doses for the study medications are: carbamazepine-600 mg., gabapentin-1500 mg., and lamotrigine-150 mg. Patients are assessed biweekly during the first 8 weeks, every 4 weeks until week 24 and every 8 weeks until week 52. Patients wishing to continue on their study drug after 52 weeks are seen quarterly for an additional year.

RESULTS: For the primary outcome measure of retention at 12 months, there was a statistically significant (p=0.0002) overall difference between the treatment groups (lamotrigine=55.8%, gabapentin=49.0%, and carbamazepine=35.5%). The paired comparisons indicated significant differences between lamotrigine and carbamazepine (p<0.0001) and gabapentin and carbamazepine (p=0.008). Consideration of reasons for early terminations indicates significant overall differences (p=0.001) between treatment groups for early terminations due to adverse events (lamotrigine=12.1%, gabapentin=21.6%, and carbamazepine=31.0%. There were significant paired comparisons for lamotrigine vs carbamazepine (p<0.0001) and lamotrigine vs gabapentin (p=0.015). There were no differences between the treatment groups for percent of patients seizure free at 3, 6, and 12 months or for the time to first, second, fifth, or tenth seizure (all p>0.05). When individual adverse events during the first 12 months on study drug were considered, it was seen that more gabapentin patients had significantly more weight gain, severe weight gain (>18 pounds), and water retention than patients on either lamotrigine or carbamazepine. Hypersensitivity (rash of any degree) occurred more frequently with carbamazpine than with lamotrigine (p=0.007). The overall conclusion is that lamotrigine and gabapentin should be considered as initial therapy for older patients with newly diagnosed seizures.

Rowan, A.J., Ramsay, R.E., Collins, J.F., Pryor, F., Boardman, K.D., Uthman, B.M., Spitz, M., Frederick, T., Towne, A., Carter, G.S., Marks, W., Felicetta, J., Tomyanovich, M.L., and the VA Cooperative Study 428 Group - New onset geriatric epilepsy. A randomized study of gabapentin, lamotrigine, and carbamazepine. Neurology 64 1868-1873, 2005

ELIGIBILITY:
Veterans 60 years of age or older who have new onset, unprovoked seizures of focal onset, with or without secondary generalization.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720
Dates: Start 1998-01; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Vamc - West Los Angeles, Los Angeles, Ca, Los Angeles, California
  - Vamc - San Diego, San Diego, Ca, San Diego, California
  - San Francisco VAMC, San Francisco, California
  - Denver VA Medical Center, Denver, Colorado
  - Vamc - Bay Pines, Fl, Bay Pines, Florida
  - Gainesville VA Medical Center, Gainesville, Florida
  - Miami VA Medical Center, Miami, Florida
  - Study Chairperson, Miami, Florida
  - Chicago VA Medical Center (West Side), Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - New Orleans VAMC, New Orleans, Louisiana
  - Boston VA Medical Center, Boston, Massachusetts
  - Bronx VA Medical Center, The Bronx, New York
  - Study Chairman, The Bronx, New York
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma
  - Vamc - Pittsburgh, Pittsburgh, Pa, Pittsburgh, Pennsylvania
  - Dallas VA Medical Center, Dallas, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia